CLINICAL TRIAL: NCT04866615
Title: Posterior Segment Evaluation of Patients With Systemic Lupus Erythematosus Using Optical Coherence Tomography and Optical Coherence Tomography Angiography
Brief Title: Posterior Segment Evaluation of Patients With SLE Using OCT and OCTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hazem Mohamed Mohamed, Principal Investigator, Minia University
Other Study IDs: OCT&OCTA in SLE
Record Dates: First submitted 2021-04-13; First posted 2021-04-30 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: SLE (Systemic Lupus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 50 patients newly diagnosed SLE with no treatment: OCT & OCTA for newly diagnosed SLE patients
  Interventions: Diagnostic Test: Optvue OCT
- 50 patients SLE on treatment by (HCQ) at doses of less than 6.5 mg/kg per day for less than 5 years: OCT & OCTA for on treatment SLE patients
  Interventions: Diagnostic Test: Optvue OCT
- 50 normal subjects as control group of similar age and gender: OCT & OCTA for normal subjects
  Interventions: Diagnostic Test: Optvue OCT

INTERVENTIONS:
Diagnostic Test: Optvue OCT — Optical coherence tomography

SUMMARY:
Aim of The Study To evaluate different structural retinal changes using OCT and OCT-A in patients with SLE ; newly diagnosed patients and patients on treatment and compare parameters with normal subjects

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune inflammatory

disease that involves different organs and systems. The heterogeneous nature of

the disease represents a great challenge in its diagnosis and management. Studies

reported that the percentage of SLE patients demonstrating ocular manifestations

can reach up to 30%.

The pathogenesis of the ocular involvement is still unclear, but immune

complex vasculopathy and inflammatory mediators might be implicated. The most

common ocular manifestation in SLE was found to be kerato-conjunctivitis

sicca(KCS) followed by retinopathy, where is the most severe manifestation was

the optic nerve involvement, which might end up with irreversible blindness while

anterior uveitis is a rare manifestation in SLE.

Retinal involvement can vary from subclinical vascular changes to vaso-

occlusive vision-threatening retinopathy. Lupus retinopathy is secondary to IgG

complex-mediated micro-angiopathy that leads to small vessels infarcts. Currently,

there is no agreement on existing biomarkers to identify SLE patients who have

subclinical retinal involvement, or to identify whether micro-vascular changes in

the retina are attributable to SLE. Lupus retinopathy is usually associated with

high disease activity especially nephritis and cerebritis.

On the other side, hydroxychloroquine,(HCQ) a cornerstone in lupus treatment, rarely causes ocular toxicity at doses of less than 6.5 mg/kg per day. Moreover, HCQ is found to be associated with retinopathy after a prolonged time of treatment (>5 years).

HCQ binds to melanin pigments in the retinal pigment epithelium (RPE). This binding may serve to concentrate the agents in the cell and contribute to their long-term effects. The classic pattern of retinal toxicity of HCQ is RPE depigmentation with foveal sparing, known as bull's-eye maculopathy. Although visual acuity in these patients seems intact, patients complain from para-central scotomas associated with reading difficulties. Besides, reduced color perception can be seen as retinopathy symptoms. That is why it is important to evaluate the eyes before starting therapy and during follow-up visits.

Modern imaging techniques have provided easier and more accurate evaluation as Optical coherence tomography (OCT) is a noninvasive imaging technology, which picks up cross-sectional pictures of the retinal layers, detect thinning of retinal nerve fiber layer and macula.

Optical coherence tomography angiography (OCTA) is a relatively new technique that allows visualization of the retina capillary bed and its subtle changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Patients with SLE diagnosed by a Rheumatologist with no ocular involvement upon clinical examination

Exclusion Criteria:

1. Patients with history of intraocular surgery as cataract surgery retinal detachment surgery and anti-glaucoma surgery.
2. Patients with significant media opacity as corneal opacity, cataract.
3. Patients with ocular diseases as glaucoma, uveitis.
4. Patients with any retinal affection as pathological myopia, macular hole, age related macular degeneration and retinal vascular occlusion.
5. Patients with systemic diseases as diabetes mellitus (DM), hypertension, abnormal kidney functions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Minia Governorate diagnosed with SLE and healthy one
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of vessel density | 3 months
  comparison of vessel density of superficial and deep layers of retina in 150 subjects divided into 3 groups newly diagnosed SLE patients and SLE patients on treatment and normal subjects using OCT Angiography.
Measurement of foveal avascular zone | 3 months
  1) comparison of foveal avascular zone between 3 groups using OCT Angiography.
Measurement of macular thickness | 3 months
  comparison of macular thickness between 3 groups using OCT.
Measurement thickness of retinal nerve fiber layer | 3 months
  Comparison of thickness of retinal nerve fiber layer between the 3 groups using OCT.
Measurement of thickness of ganglion cell layer complex | 3 months
  Comparison of thickness of ganglion cell layer complex between the 3 groups using OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Shehab, MD, Study Director — Minia University Hospital; Mohamed Farouk, MD, Study Director — Minia University Hospital; Mohamed Salah, MD, Study Director — Minia University Hospital; Hazem Mohamed, Resident, Principal Investigator — Minia University Hospital
Locations (1):
- Minia university hospital, Minya, Egypt

REFERENCES:
- [Background] Larosa M, Iaccarino L, Gatto M, Punzi L, Doria A. Advances in the diagnosis and classification of systemic lupus erythematosus. Expert Rev Clin Immunol. 2016 Dec;12(12):1309-1320. doi: 10.1080/1744666X.2016.1206470. Epub 2016 Jul 8. PMID 27362864
- [Background] Shoughy SS, Tabbara KF. Ocular findings in systemic lupus erythematosus. Saudi J Ophthalmol. 2016 Apr-Jun;30(2):117-21. doi: 10.1016/j.sjopt.2016.02.001. Epub 2016 Feb 16. PMID 27330388
- [Background] El-Shereef RR, Mohamed AS, Hamdy L. Ocular manifestation of systemic lupus erythematosus. Rheumatol Int. 2013 Jun;33(6):1637-42. doi: 10.1007/s00296-011-2296-x. Epub 2011 Dec 28. PMID 22202921
- [Background] Kahwage PP, Ferriani MP, Furtado JM, de Carvalho LM, Pileggi GS, Gomes FH, Terreri MT, Magalhaes CS, Pereira RM, Sacchetti SB, Marini R, Bonfa E, Silva CA, Ferriani VP. Uveitis in childhood-onset systemic lupus erythematosus patients: a multicenter survey. Clin Rheumatol. 2017 Mar;36(3):547-553. doi: 10.1007/s10067-016-3534-0. Epub 2017 Jan 9. PMID 28070763
- [Background] Sivaraj RR, Durrani OM, Denniston AK, Murray PI, Gordon C. Ocular manifestations of systemic lupus erythematosus. Rheumatology (Oxford). 2007 Dec;46(12):1757-62. doi: 10.1093/rheumatology/kem173. Epub 2007 Aug 5. PMID 17681981
- [Background] Farrell DF. Retinal toxicity to antimalarial drugs: chloroquine and hydroxychloroquine: a neurophysiologic study. Clin Ophthalmol. 2012;6:377-83. doi: 10.2147/OPTH.S27731. Epub 2012 Mar 8. PMID 22457587
- [Background] Marmor MF, Kellner U, Lai TY, Melles RB, Mieler WF; American Academy of Ophthalmology. Recommendations on Screening for Chloroquine and Hydroxychloroquine Retinopathy (2016 Revision). Ophthalmology. 2016 Jun;123(6):1386-94. doi: 10.1016/j.ophtha.2016.01.058. Epub 2016 Mar 16. PMID 26992838